CLINICAL TRIAL: NCT01242254
Title: An Open Label, Multicenter, Randomized, Uncontrolled Study Assessing the Safety and Efficacy of KH902 in Patients With Choroidal Neovascularization Due to Neovascular Age-related Macular Degeneration(HOPE Study)
Brief Title: A Study Assessing the Safety and Efficacy of Multiple Intravitreal KH902 in Patients With CNV Due to AMD
Acronym: HOPE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Collaborators: University of Wisconsin, Madison (Other); Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHSWKH902004
Record Dates: First submitted 2010-11-10; First posted 2010-11-16 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2011-07

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: KH902; age-related macular degeneration; choroidal neovascularization; intravitreal injection; multiple injections
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Patients will receive an intravitreal injection of KH902 0.5mg/eye/time monthly, after 3-time treatment patients will go on an as needed (PRN) dosing phase till week 52
  Interventions: Biological: Intravitreal injection of KH902
- Group B (Experimental): Patients will receive an intravitreal injection of KH902 2.0mg/eye/time monthly, after 3-time treatment patients will go on an as needed (PRN) dosing phase till week 52
  Interventions: Biological: Intravitreal injection of KH902

INTERVENTIONS:
Biological: Intravitreal injection of KH902 — 0.5 mg 2.0 mg once per 4 weeks during fixed dosing phase once as needed during extended treatment phase

SUMMARY:
This study is designed to assess the efficacy and safety of multiple intravitreal injection of KH902 in patients with CNV due to AMD.

DETAILED DESCRIPTION:
Due to conclusions of KH902 Ia study:

Doses of single intravitreal injection of a recombinant human VEGF receptor-Fc fusion protein (KH902) in patients with CNV secondary to neovascular AMD are from 0.05 mg to 3.0 mg. The trial shows that KH902 is safe and tolerable, and no DLT, ophthalmia reaction, endophthalmitis, or systemic AE relevant to the drug is reported, and the main AEs are transient ocular tension increase and micro-hemorrhage in injection site. KH902 appears to produce rapid clinical effects on VA, supported by improvements in anatomical features, in patients with neovascular AMD.

HOPE Study is an open label, multi-center, randomized, uncontrolled dose-and interval-ranging phase Ib study designed to assess the efficacy and safety of multiple intravitreal injection of KH902 at variable dosing regimen in patients with CNV due to AMD. Two groups of patients will initially receive intravitreal administration of KH902 following the randomization:

1. Patients in group A will receive monthly intravitreal injections of KH902 for 3 times successively at a dose of 0.5 mg/50 μl/eye;
2. Patients in group B will receive monthly intravitreal injections of KH902 for 3 times successively at a dose of 2.0 mg/50 μl/eye.

Following the initial 12-week fixed-dosing phase of the trial:

Patients in group A and group B will continue to receive monthly intravitreal injections of KH902 with 0.5 mg/50 μl/eye or 2.0 mg/50 μl/eye as same as the doses he/she received during the fixed dosing phase, on an as needed (PRN) dosing schedule, based upon the need for re-treatment in accordance with pre-specified criteria up till week 52.

ELIGIBILITY:
Inclusion Criteria:

* Signed the Informed Consent Form by patients or legal representative;
* Men and women ≥ 45 years of age;
* Active primary or recurrent lesions with CNV secondary to neovascular AMD;
* Total lesion size ≤ 12 disc areas in either eye;
* BCVA of the study eyes < 69 letters and the BCVA of fellow eyes ≥ 19 letters;
* Clear ocular media and adequate pupil dilation.

Exclusion Criteria:

* CNV lesion secondary to ocular conditions other than neovascular AMD
* History of vitreous hemorrhage, retinal tear, rhegmatogenous retinal detachment or macular hole in the study eye;
* Presence of retinal detachment, retinal pigment epithelial tear, or retinal macular traction in the study eye;
* Anaphylactic disease;
* Uncontrolled glaucoma in either eye;
* Current active ocular inflammation or infection in either eye;
* Previous anti-VEGF drug treatment in the study eye within three months preceding screening, and/or, for the fellow eye, within one month preceding screening;
* Previous ophthalmologic operation or laser therapy in the study eye within three months preceding screening;
* Current non-healing wound, ulcer, fractures, etc;
* Uncontrolled systemic conditions;
* Patients of child-bearing potential do not adopted adequate contraception methods;
* Pregnant or nursing women.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The incidence rate of adverse event | at 52 week
  To evaluate the safety of multiple intravitreal injection of KH902 of each group.

SECONDARY OUTCOMES:
Change from Baseline in BCVA | Specified timepoints during the screening phase and 52-week treatment period
  To evaluate the efficacy of multiple intravitreal injection of KH902 of each group in the mean change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Junjun Zhang, Principal Investigator — West China Hospital
Locations (3):
- China (3):
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital ,Sichuan University, Chengdu, Sichuan